# CONFIDENTIAL FORM STATISTICAL ANALYSIS PLAN N° DGD-55-003 VERSION N° 2 DATED: 26 FEBRUARY 2018 (REF 1011622) F015830-01 F0age 1 / 49

# STATISTICAL ANALYSIS PLAN No DGD-55-003

#### THE NSsaFe STUDY

Observational Study on the incidence of NSF in renal impaired patients following  $DOTAREM^{\text{\scriptsize \$}}\ administration$ 

| SPONSOR | STATISTICAL ANALYSIS PLAN |
|-------------------------------------------|---------------------------|
| GUERBET | APPROVAL |
| B.P. 57400 | |
| 95943 ROISSY CHARLES DE GAULLE CEDEX - | |
| FRANCE | |
| T. 1. 22 1.45 01.5000 | |
| Tel.: 33-1-45-91-5000 | |
| Fax: 33-1-45-91-5199 | |
| BIOSTATISTICIAN | Date and Visa |
| Florence Praud | Dute and Visa |
| Troine Trad | |
| Tel. 33-1-85-65-7735 | |
| e-mail: fpraud@inferential.fr | |
| DIOCT ATTICTICIAN | D 4 IV |
| BIOSTATISTICIAN | Date and Visa |
| Benoit PIEDNOIR | |
| Tel. 33-1-45-91-4642 | |
| e-mail: benoit.piednoir@guerbet-group.com | |
| <u> </u> | |

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

# **HISTORY FORM**

| Version | Date | Statistician | Reason for change |
|---------|------------------|-----------------|-------------------|
| 1.0 | 12 october 2017 | Benoit PIEDNOIR | Initial Version |
| 2.0 | 26 february 2018 | Florence PRAUD | Implementation of |
| | | | comments on 1.0 |

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

# LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

AE Adverse Event BMI Body Mass Index

GBCA Gadolinium based Contrast Agent

DRM Data Review Meeting

eGFR Estimated Glomerular Filtration Rate

MedDRA Medical Dictionary For Regulatory Activities

MR Magnetic Resonance

MRI Magnetic Resonance Imaging NSF Nephrogenic Systemic Fibrosis

PT Preferred Term

SAE Serious Adverse Event SD Standard Deviation SOC System Organ Class

TEAE Treatment Emergent Adverse Event

# CONFIDENTIAL

#### **FORM**

# F015830-01

# STATISTICAL ANALYSIS PLAN N° DGD-55-003

VERSION N° 2

DATED: 26 FEBRUARY 2018

Page 4 / 49

# (REF 1011622)

#### **TABLE OF CONTENTS**

| нізт | UKY FURM | |
|---|---|---|
| LIST ( | OF ABBREVIATIONS AND DEFINITION OF TERMS | 3 |
| 1. St | UMMARY OF THE STUDY PROTOCOL | 6 |
| 1.1. | STUDY OBJECTIVES | 6 |
| 1.2. | | |
| 1.3. | STUDY CONTRAST MEDIA | 7 |
| 2. E | VALUATION CRITERIA | 8 |
| 2.1. | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 8 |
| 2.2. | Efficacy criteria | 8 |
| 2.3. | | |
| 2.4. | | _ |
| 3. S | TATISTICAL METHODS | 10 |
| 3.1. | | |
| 3.2. | | |
| 3.3. | | |
| 3.4. | | |
| 3.5.<br>3.6. | | |
| 3.7. | | |
| 3.8. | | |
| 3.9. | | |
| 3.10 | ). ACTIVE CONTROL STUDIES INTENDED TO SHOW EQUIVALENCE | 11 |
| 3.11 | EXAMINATIONS OF SUBGROUPS | 11 |
| 4. C | CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES | 12 |
| 5. S | TATISTICAL AND ANALYTICAL PLANS | 13 |
| 5.1. | DISPOSITION OF SUBJECTS | 13 |
| 5.2. | | |
| 5.3. | MEASUREMENTS OF STUDY DRUG COMPLIANCE | |
| 5.4. | | |
| 5.5. | | |
| 5.6. | | |
| | .6.1. Extent of Exposure | |
| | .6.3. Adverse Events | |
| | .6.4. Deaths, serious adverse events and other significant adverse events | |
| | .6.5. Clinical laboratory evaluation | |
| | .6.6. Vital signs, physical findings and other observations related to safety | |
| 6. L | IST OF TABLES, FIGURES AND LISTINGS | 20 |
| 6.1. | | |
| 6.2. | | 20 |
| 6. | .2.1. Demographic Data Summary and Figures | 20 |
| | .2.2. Efficacy Data Summary Figures and Tables | 21 |
| | .2.3. Safety Data Summary Figures and Tables | 21 |
| 6.3. | | |
| 6. | .3.1. Disposition of Subjects | 22 |

# CONFIDENTIAL FORM STATISTICAL ANALYSIS PLAN N° DGD-55-003 VERSION N° 2 DATED: 26 FEBRUARY 2018 (REF 1011622) F015830-01 Page 5 / 49

| Q A | PPFNDICES | 40 |
|---|---|---|
| 8. R | EFERENCES | 48 |
| 7.3. | CONTENTS OF CLINICAL STUDY REPORT SECTION 16.2 | 41 |
| 7.2. | | |
| 7.1. | CLINICAL STUDY REPORT IN-TEXT TABLES, FIGURES AND LISTINGS | 24 |
| 7. SI | HELLS FOR TABLES, FIGURES AND LISTINGS | 24 |
| 6 | 3.9. Vital signs, Physical Findings and Other Observations Related to Safety | 23 |
| 6 | 3.8. Listing of Individual Laboratory Measurements | |
| 6 | 3.7. Adverse Event Listings | |
| 6 | 3.6. Individual Efficacy Response Data | |
| 6 | 3.5. Compliance and/or Drug Concentration Data | |
| 6 | 3.4. Demographic Data and Baseline Characteristics | |
| 6 | 3.3. Subjects Excluded from Efficacy Analysis | |
| 6 | 3.2. Protocol Deviations | |

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

#### 1. SUMMARY OF THE STUDY PROTOCOL

This document presents the statistical analysis plan (SAP) for Guerbet, Protocol No. DGD-55-003: "Observational study on the incidence of NSF in renal impaired patients following DOTAREM® administration".

This analysis plan is based on the final protocol Version 1.0 dated November 08, 2010 + protocol amendment 1 dated July 24, 2012.

# 1.1. Study objectives

The primary objective of this study is to prospectively estimate the incidence of NSF in patients with moderate to severe renal impairment after administration of DOTAREM®. Patients will be followed during a two-year period after administration of DOTAREM®, to assess if signs or symptoms suggestive of NSF have appeared.

The secondary objectives of the study are:

- to collect a large number of data concerning the general safety profile of DOTAREM® during patient inclusion and MR examination,
- to collect information regarding MRI indication,
- to collect conditions of use/administration of the product in this specific population of patients,
- to collect efficacy data (image and diagnostic quality).

#### 1.2. Study design

DGD-55-003 is a prospective multinational, multicenter, observational Post-Marketing Study (PMS) including longitudinal safety follow-ups. The number of sites and patients will vary from one country to another.

Patients included in the study should have moderate (eGFR of 30-59 ml/min/1.73 m²) to severe (eGFR<30 ml/min/1.73 m²) and end stage (eGFR<15 ml/min/1.73 m²) renal impairment or dialysis and should be scheduled for a contrast-enhanced MRI with DOTAREM®.

After a patient has satisfied all eligibility requirements, he will undergo a MRI examination with a DOTAREM® administration. All patients will be followed up during 2 years after DOTAREM® administration to collect data on any suspected NSF or NSF related symptoms.

The images will be assessed on-site by the same investigator at each participating hospital.

Safety assessments will include adverse events that occurred during the MRI examination or during the time of usual follow-up post DOTAREM® administration.

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

# 1.3. Study contrast media

DOTAREM® (gadoterate meglumine)

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

#### 2. EVALUATION CRITERIA

# 2.1. Demographic and other baseline characteristics

Demographic variables collected for this study are:

- Age in years for patient more than 2 years old and age in months otherwise,
- height,
- weight,
- sex.

Baseline characteristics collected for this study are:

- Magnetic field,
- Current renal status according to the investigator,
- Most recent serum creatinine before inclusion (in mg/L or mg/dL or μmol/L),
- Estimated creatinine clearance for children less than 2 years old and eGFR otherwise,
- Pre-existing risk factors and medical history,
- Previous examinations with GBCA,
- Concomitant treatment and recent surgery (<2 years),
- Indication of MRI examination,
- Premedication.

#### 2.2. Efficacy criteria

The primary objective of the study is related to the NSF prevalence and therefore the primary criterion is not an efficacy criterion.

Efficacy variables are derived from the investigator evaluations of the imaging examination. Images will be rated regarding the following items:

- Image quality
- Diagnostic quality

### 2.3. Safety criteria

Safety variables collected for this study are:

- Modalities of DOTAREM® administration
  - o Volume injected,
  - o Type of injection,
  - o Number of injections,
  - Nature of package
- From DOTAREM® administration until end of usual follow up in the MR unit
  - o Adverse events,
  - Serious adverse events,
  - o Adverse events requiring the administration of a concomitant drug,
  - o Adverse events according to intensity and outcome,
  - o Adverse events related to contrast media injection.
- During the follow-up period

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

- o Suspicion of NSF and final diagnosis of NSF,
- o Medical events,
- o Serum creatinine measurements.

# 2.4. Other criteria

None

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

#### 3. STATISTICAL METHODS

#### 3.1. General considerations

At the end of the study, after the database lock, the statistical analysis will be performed by GUERBET Biostatistic team on the basis of the present document.

A quality control of the statistical analysis will be performed to ensure the reliability of the results.

Thorough description of all parameters reported will be presented. Summary tabulated results will be provided by assessment time if relevant or they will be replaced by the corresponding individual data listings if too few patients are concerned.

Tabulations of quantitative parameters will include the following summary statistics: Number of Patients / Mean / Standard Deviation / Minimum / Median / Maximum. If for a given parameter, the raw value has been collected with x decimal places, the mean, median and standard deviation will be rounded to x+1 decimal places, while the minimum and maximum values will be tabulated as reported with x decimal places.

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category as well as the percentage (%). Percentages will be rounded to one decimal place. The category missing will be displayed only if there are actually missing values. Percentages will be calculated on the total of recorded (non missing) data.

The **baseline value** will be defined as the last available value prior to administration of the investigational product.

No statistical tests will be performed in this study. All statistics will be only descriptive.

SAS® Version: 9.4 will be used for all descriptive summaries.

# 3.2. Null and alternative hypothesis

None as no statistical test will be performed in this study.

#### 3.3. Determination of sample size

This study aims at accurately estimating the incidence of the NSF in renal impaired patients, in case such an event is observed after injection of DOTAREM®. Assuming that when exposed to GBCA, the frequency of NSF is ranging from 0% to 4% in this population (maximum frequency being observed with linear GBCA), with a sample size of 1000 patients, a two-sided 95% exact confidence interval for a single proportion will allow to estimate with an adequate accuracy the frequency of this event according to the following table:

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

| | | Observed | |
|----------------|------|-----------|---------------|
| Observed cases | N | frequency | Exact 95% IC |
| 0 | 1000 | 0.0% | 0.00% - 0.37% |
| 1 | 1000 | 0.1% | 0.00% - 0.56% |
| 2 | 1000 | 0.2% | 0.02% - 0.72% |
| 5 | 1000 | 0.5% | 0.16% - 1.16% |
| 10 | 1000 | 1.0% | 0.48% - 1.83% |
| 15 | 1000 | 1.5% | 0.84% - 2.46% |
| 20 | 1000 | 2.0% | 1.23% - 3.07% |
| 30 | 1000 | 3.0% | 2.03% - 4.26% |

The sample size of 1000 patients was not reached before the end of the enrolment period (see section 4)

# 3.4. Adjustment for covariates

Not applicable

#### 3.5. Handling of dropouts or missing data

If the start date of an adverse event is missing, then the adverse event occurs after the DOTAREM® injection.

No replacement of missing data is planned in this study.

#### 3.6. Interim analyses and data monitoring

Not applicable

#### 3.7. Multicentre studies

Number of patients included in each centre will be presented but no demographic parameters, baseline characteristics, efficacy or safety criteria will be presented by centre.

#### 3.8. Multiple comparisons/Multiplicity

Not applicable

# 3.9. Use of an "efficacy subset" of patients

Efficacy results will be presented using the set of patients having an available diagnostic assessment.

# 3.10. Active control studies intended to show equivalence

Not applicable

#### 3.11. Examinations of subgroups

Not applicable

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

#### 4. CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES

The protocol was amended on one occurrence globally and twice in Turkey and twice in the United State of America (see protocol amendments for a full list of changes).

The global amendment has introduced following changes:

- The minimum number of patients with severe renal impairment was changed from 50% to 40% but this does not change the planned analysis as no analysis is foreseen considering the renal impairment status.
- The period of recruitment was extended. Initially 1000 patients were supposed to be included in the study with a minimum of 50% of patients with severe renal impairment. Despite the extension of the recruitment period, the sample size of 1000 patients was not reached by the end of the recruitment period. Thanks to better understanding of causality and risk factors conducting to NSF occurrence, safety and educational measures starting from 2012, the rate of NSF appears to be less than 1%, and the study was no longer powered to assess the NSF rate. For this reason and taken into account that the NSF was not a safety priority for the competent authorities anymore due to the low incidence, the recruitment was stopped in March 2015.
- Patients who had received DOTAREM® within 12 months prior to inclusion were included in the study.

The methodology of statistical testing is described in the protocol although no comparison is possible. No statistical tests will be presented in the report.

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

#### 5. STATISTICAL AND ANALYTICAL PLANS

#### 5.1. Disposition of patients

Patient disposition will be based on all included patients (that is to say patients included in the study by having a questionnaire partly or fully filled in) and will display patients prematurely withdrawn of the study and reasons why patients were prematurely withdrawn.

Frequency of patients by centre within country and frequency of patients by visits will be tabulated. Amongst patients indicated as having undergone the follow-up, some were indicated as being prematurely withdrawn from the study. These patients had either no results collected at this visit or only one result (no suspicion of NSF), therefore it has been decided that the reliable data is the withdrawal form and so these patients were eventually considered as having not undergone the follow-up 3 visit.

Centre characteristics and radiological activities of centres will be tabulated.

A listing showing disposition of patients and a listing showing centre characteristics and radiological activities of centres will be provided in CSR appendix 16.2.1.

#### 5.2. Data Sets Analysed and protocol deviations

#### Data sets analysed

There will be three patient populations defined for this study: all-included population (AIP), safety population (SP) and efficacy population (EP).

The all-included population (AIP) will include all patients who have a questionnaire partly or fully filled in. This population will be used for the description of disposition of patients, protocol deviations and demographic data.

The safety population (SP) will include all patients receiving at least one injection of contrast media regardless of the quantity. This population will be used to evaluate the NSF occurrence, to describe administration modalities, for analysis of adverse events, laboratory data, other safety observations, medical events and concomitant medications presentation. Furthermore, demographic data and medical history will be presented using this population as well.

The efficacy population (EP) will include all patients who have an available imaging assessment.

The following table describes how the above-defined patients populations will be used in the different analyses conducted.

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

Analysed populations

| Analysed Populations | AIP | SP | EP |
|---|---|---|---|
| Population characteristics | ✓(only Demographics) | ✓ | |
| Exposure | | ✓ | |
| Efficacy assessment | | | ✓ |
| Safety assessment: Main criterion | | ✓ | |
| Safety assessment: Secondary criteria (AE, laboratory data and other safety observation) | | ✓ | |
| Concomitant medications | | ✓ | |

Frequency and percentages of patients in each population will be presented. A listing showing the distribution of each patient in the populations will also be provided in CSR appendix 16.2.3.

#### Protocol deviations

A protocol deviation is any change, divergence, or departure from the study design or procedures defined in the protocol that might significantly affect the completeness, accuracy, and/or reliability of the study data or that might significantly affect a patient's rights, safety, or well-being. Protocol deviations are to be displayed in the Clinical Study Report (CSR) as a metric of the feasibility and reliability of the study.

The list of protocol deviations is defined in this document but protocol deviations can be added during the Data Review Meeting (DRM). Protocol deviations will be extensively sought from, clinical database and monitoring files (if monitoring was required as per local regulation).

As no efficacy or safety subset are defined, no deviation will lead to exclusion from this subset and therefore deviations will not be split in major and non major deviations.

The deviations are listed in the table below:

| Category | Description |
|---|---|
| Inclusion/Non-inclusion | Patient <b>not</b> scheduled for a contrast enhanced MRI with DOTAREM® |
| criteria not met | or who will not be followed up for his/her renal impairment by one of |
| | the site study co-investigators |
| | Patient having mild renal impairment (eGFR 60-89 mL/min/1.73 m <sup>2</sup> ) |
| | or normal renal function (eGFR>90 mL/min/1.73 m <sup>2</sup> ) |
| | Patient has received a GBCA other than DOTAREM® within the past |
| | 12 months prior to inclusion in this study |
| | Patient has experienced a previous hypersensitivity reaction to GBCA |
| Non respect of study | Patient is not injected |
| schedule and procedures | |
| | Follow-up 1 visit is not performed |

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

| Follow-up 2 visit is not performed |
|------------------------------------------------------------------------|
| Follow-up 3 visit is not performed |
| Follow-up 1 visit is not done between 3 and 12 months after the study |
| drug administration |
| Follow-up 2 visit is not done between 13 and 21 months after the study |
| drug administration |
| Follow-up 1 visit is not done between 22 and 27 months after the study |
| drug administration |
| The interval of at least 3 months was not respected between two |
| follow-up visits. |

No deviation will lead to exclusion from analyses in this safety study.

#### 5.3. Measurements of study drug compliance

None

#### 5.4. Demographic and Other Baseline Characteristics

All demographic variables and other baseline characteristics will be presented using the SP. Demographics variables will be presented using the AIP as well.

#### **Demography**

Summary statistics for quantitative variable will be calculated for age, body weight, height and BMI. Frequency and percentages will be calculated for gender.

BMI will be derived for each collection of body weight using the formula:  $BMI = \frac{BodyWeight_{(Kg)}}{Height_{(m)}^2}$ 

#### **Magnetic Field**

Summary statistics for qualitative variable will be presented for magnetic field (in tesla).

#### **Current renal status**

Summary statistics for quantitative variable will be calculated for serum creatinine, estimated creatinine clearance and eGFR. Frequency and percentages will be calculated for current renal status.

Serum creatinine will be presented in  $\mu$ mol/L. Therefore, conversion will apply for measurement in mg/L and mg/dL using the following conversion factors [1]:

From mg/dL to µmol/L: multiply by 88.4 From mg/L to µmol/L: multiply by 8.84

Should be noted that an aberrant result of serum creatinine was entered in the database for one patient (1.36  $\mu$ mol/L). As it was impossible to correct this discrepancy in the database, it was decided not to present it in the statistical results of the clinical study report.

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

The estimated creatinine clearance (mL/min) will be calculated using the Schwartz formula for children less than 2 years old. The eGFR (mL/min/1.73 m²) will be calculated using the MDRD formula otherwise. They will be presented independently.

#### Risk factors

Frequency and percentages will be calculated for each risk factor. Specification for other cardiovascular disease, nervous system disorders, other treatments at risk and dose of Erythropoietin will be only listed.

#### Previous examination with GBCA

Number of patients with at least one previous examination with GBCA will be displayed globally and by classified name of product. Name of product will be classified as the following:

- If the words "Gadovist" or "Gadavist" appear in the product name then class=" Gadobutrol"
- If the word "Dotarem" appears in the product name then class= "Gadoterate meglumine"
- If the word "Primovist" or "Gd-EOB-DTPA" or "Gd EOB" appear in the product name then class= "Gadotexate disodium"
- If the words "Magnevist" or "Gadopentetate" appear in the product name then class= "Gadopentetate dimeglumine"
- If the word "Multihance" appears in the product name then class= "Gadobenic acid meglumine"
- If the word "Omniscan" appears in the product name then class= "Gadodiamide"
- If the word "Optimark" appears in the product name then class="Gadoversetamide"
- If the words "No contrast" or "without contrast" or "NA" or "Non-contrast brain MRI" appear in the product name then class = "Without Contrast"
- If the words "Unknown" or "MD" or "UN" or nothing appear in the product name then class = "Missing"
- Otherwise then class="Other"

#### **Recent surgeries**

Surgeries done less than two years before the MRI examination with DOTAREM® will be only listed. Number of patients with at least one surgery will be tabulated.

#### **Concomitant treatments**

Concomitant treatments at the time of the MRI examination with DOTAREM® will only be listed. Number of patients with at least one concomitant medication will be tabulated.

#### **Indication of MRI examination**

Indication of MRI examination will be tabulated by main classification (Central nervous system, whole body, musculoskeletal system, angiography and other) and sub classification.

Some indications for MRI categorized as "Other" should be classified in pre-defined categories according to the following algorithm:

If the wording contains "angio" or "anjio" then classify to Angiography system and according to the following for the sub classification:

| If the wording is: | Specified Organ |
|--------------------------------------------------|-----------------|
| "kidney" or "kidneys" or "renal" or contains one | 2=Renal |
| of these | |

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

| "iliac" or contains "iliac" | 3=Aorto iliac |
|-----------------------------|---------------|
| "calf" | 4=Calf |
| "Otherwise" | 5=Other |

Otherwise classify to whole body system and according to the following. for the sub classification:

| If the wording is: | Specified Organ |
|----------------------------------------------------|-----------------|
| "liver" or contains "lilver" | 1=Liver |
| "kidney" or "kidneys" or "renal" or contains one | 2=Kidney |
| of these | |
| "pancreas" | 3=Pancreas |
| "pelvis" or contains "pelvic" or contains "pelvin" | 4=Pelvis |
| "lung" | 5=Lung |
| "heart" or "cardiac" or "cardio" | 6=Heart |
| "breast" | 7=Breast |

#### Premedication

Patients having received at least one premedication will be presented. Premedication received will be only listed.

Listings of all demographic parameters and baseline characteristics will be presented in CSR Appendix 16.2.4.

#### 5.5. Efficacy evaluation

All efficacy analyses will be conducted using the EP.

#### Image quality

Frequency of images with very poor, poor, fair, good and very good quality will be presented.

# Diagnostic quality

Diagnosis assessment (Yes/No) and reason for impossible diagnosis will be tabulated. Diagnosis when available will be listed.

Listing of all efficacy data will be presented in CSR appendix 16.2.6.

#### 5.6. Safety Evaluation

All safety analyses will be conducted using the SP.

#### 5.6.1. Extent of Exposure

Extent of exposure will present the DOTAREM® administration: total volume injected, type of injection, number of injections (1 or 2), nature of package, and volume of vial and pre-filled syringe used. Total dose injected (mL/kg), calculated by dividing the total volume of DOTAREM® administered by the body weight will be presented as well.

Summary statistics for quantitative variable will be calculated for total volume injected and total dose injected. Frequency and percentages will be calculated for other criteria.

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

Listing of exposure will be presented in CSR appendix 16.2.5.

# 5.6.2. Primary safety endpoint: NSF

The number and percentage of patients with any suspicion of NSF will be presented.

For patients having any suspicion of NSF, the reasons of the suspicion will be tabulated

Among patient having any suspicion of NSF, the number and percentage of patients with a confirmatory biopsy or not (and the reason if not) will be presented.

Among patients having a confirmatory biopsy, the number and percentage of patients with a final diagnosis of NSF or not (and the reason if not) will be presented.

Listing of NSF suspicion and diagnosis will be presented in CSR appendix 16.2.9.1

#### 5.6.3. Adverse Events

Adverse events (AEs) will be coded in system organ classes and preferred terms using MedDRA dictionary v16.0.

Adverse events occurring or worsening after the "Treatment start date" (Date of MRI examination with DOTAREM®) will be considered as **treatment-emergent** adverse events (TEAEs).

An adverse event will be considered **related to** DOTAREM®, if the relationship to the study drug is doubtful, possible, not assessable or missing.

All AEs will be summarized in an incidence table and a specific table will focus on incidence of TEAEs.

Incidence tables will present the number and percent of patients reporting TEAEs, the number and percent of patients reporting serious adverse events (SAEs) and the number and percent of patients reporting related AEs by system organ class and preferred term.

Adverse event listings will be presented in CSR appendix 16.2.7.

#### 5.6.4. Deaths, serious adverse events and other significant adverse events

All deaths and all SAEs experienced during the study will be separately listed sorted by patient number, presenting: , emergence, diagnosis or nature, system organ class (SOC), preferred term (PT), start date, the intensity, the relationship to study drug, the outcome, the action taken and the seriousness criteria.

# 5.6.5. Clinical laboratory evaluation

Serum creatinine collected during the follow-up period will be tabulated as quantitative parameter by visit in raw data and change from baseline. If during the follow-up visits, the date of last renal function assessment is replicated then only the first measurement will be taken into account. Serum creatinine will be presented in  $\mu$ mol/L. Therefore, conversion will apply for measurement in mg/L and mg/dL using the following conversion factors [1]:

From mg/dL to  $\mu$ mol/L: multiply by 88.4 From mg/L to  $\mu$ mol/L: multiply by 8.84

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

Listing of clinical laboratory evaluation will be presented in CSR appendix 16.2.8.

# 5.6.6. Vital signs, physical findings and other observations related to safety

Medical events will be coded in body systems and preferred terms using MedDRA dictionary v16.0.

#### **Medical Event overview**

Number and percentage of patient having undergone medical events will be tabulated by follow-up visit

#### MRI examination

Number of patients with MRI examination will be displayed by follow-up visit and by name of product. Name of product will be coded using WHO DD 2015 version and will be tabulated according to ATC code.

# Medical Event by SOC and PT

Medical events will be displayed by follow-up visit and by SOC and PT.

Listing of medical events will be presented in CSR appendix 16.2.9.

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

# 6. LIST OF TABLES, FIGURES AND LISTINGS

# 6.1. Clinical study report in-text tables, figures and listings

# 6.2. Contents of clinical study report section 14

# 6.2.1. Demographic Data Summary and Figures (Section 14.1 of ICH report)

# 6.2.1.1 Disposition of Patients

| Table 14.1.1.1 | Patient Overall Disposition - All Included Population |
|---|---|
| Table 14.1.1.2 | Disposition by Visit - All Included Population |
| Table 14.1.1.3 | Disposition by Site - All Included Population |
| Table 14.1.1.4 | Centre Characteristics and Radiological Activities - All Centres |
| Table 14.1.1.5 | Magnetic Fields of MR Equipments - All MR Equipments |

#### 6.2.1.2 Protocol Deviations

Table 14.1.2.1 Protocol Deviations - All Included Population

#### 6.2.1.3 Data Set Analysed

Table 14.1.3.1 Analysis Data Populations - All Included Population

# 6.2.1.4 Demographics and Baseline Characteristics

| Table 14.1.4.1.1 | Demographic Characteristics - All Included Population |
|---|---|
| Table 14.1.4.1.2 | Demographic Characteristics – Safety Population |
| Table 14.1.4.2 | Magnetic Field – Safety Population |
| Table 14.1.4.3 | Current Renal Status - Safety Population |
| Table 14.1.4.4 | Pre-existing Risk Factor and Medical History - Safety Population |
| Table 14.1.4.5 | Previous Examinations with GBCA - Safety Population |
| Table 14.1.4.6 | Recent Surgery - Safety Population |
| Table 14.1.4.7 | Concomitant Medications - Safety Population |
| Table 14.1.4.8 | Indication of MRI Examination - Safety Population |
| Table 14.1.4.9 | Premedications - Safety Population |

|---|---|---|
| | STATISTICAL ANALYSIS PLAN N° DGD-55-003 | |
| | (REF 1011622) | |
| 6.2.2 Efficacy Data | a Summary Figures and Tables | |
| • | 4.2 of ICH report) | |
| | icacy Variables<br>2.1 of ICH report) | |
| Not applicable. | | |
| 6.2.2.2 Secondary E | Efficacy Variables | |
| Table 14.2.2.1 | Overall Quality of Images - Efficacy Population | |
| Table 14.2.2.2 | Diagnostic Quality - Efficacy Population | |
| (Section 1 | Summary Figures and Tables 4.3 of ICH report) | |
| 6.2.3.1 Extent of Ex | | |
| Table 14.3.1.1 | DOTAREM® Administration at Inclusion Visit - Safety Population | |
| - | on and diagnoses | |
| Table 14.3.2.1 Table 14.3.2.2 | Suspected NSF - Safety Population Confirmatory Biopsy and Final Diagnosis - Safety Population - | Patient with |
| | Suspicion of NSF | |
| 6.2.3.3 Displays of | Adverse Events | |
| Table 14.3.3.1 | Overall Safety Summary - Safety Population | |
| Table 14.3.3.2 | Treatment Emergent Adverse Events - Overall Summary - Safety Popula | ation |
| Table 14.3.3.3 | Pre-injection Adverse Events by Primary System Organ Class and Pref<br>Safety Population | Perred Term - |
| Table 14.3.3.4 | Treatment Emergent Adverse Events by Primary System Organ Class a<br>Term - Safety Population | and Preferred |
| Table 14.3.3.5 | Serious Treatment Emergent Adverse Events by Primary System Org<br>Preferred Term - Safety Population | an Class and |
| Table 14.3.3.6 | Treatment Emergent Adverse Events with Relationship to DOTAREM System Organ Class and Preferred Term - Safety Population | ® by Primary |
| 6.2.3.4 Listings of L | Deaths, Other Serious and Significant Adverse Events | |
| Table 14.3.3.7 | Listing of Deaths - Safety Population | |
| Table 14.3.3.8 | Listing of Serious Adverse Events - Safety Population | |

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

#### 6.2.3.5 Narratives of Deaths, Other Serious and Significant Adverse Events

Not applicable.

#### 6.2.3.6 Display of Clinical Laboratory Data

Table 14.3.4.1 Renal Status during Follow-up Period - Safety Population

#### 6.2.3.7 Vital Signs, Physical Findings and Other Observations Related to Safety

| Table 14.3.5.1 | Medical Events except MRI Examination during Follow-up Period - Safety Population |
|---|---|
| Table 14.3.5.2 | Contrast Media for MRI Examination during Follow-up Period - Safety Population |
| Table 14.3.5.3 | Medical Events except MRI Examination during Follow-up Period by Primary System Organ Class and Preferred Term - Safety Population |

# 6.3. Contents of clinical study report section 16.2

#### 6.3.1. Disposition of Patients

(Section 16.2.1 of ICH report)

| Listing 16.2.1.1 | Visit Dates - All Included Population |
|------------------|----------------------------------------------------|
| Listing 16.2.1.2 | Premature Withdrawal |
| Listing 16.2.1.3 | Centre Characteristics and Radiological Activities |

#### 6.3.2. Protocol Deviations

(Section 16.2.2 of ICH report)

Listing 16.2.2.1 Protocol Deviations - All Included Population

#### 6.3.3. Patients Excluded from Efficacy Analysis

(Section 16.2.3 of ICH report)

Listing 16.2.3.1 Analysis Data Populations - All Included Population

# 6.3.4. Demographic Data and Baseline Characteristics

(Section 16.2.4 of ICH report)

| Listing 16.2.4.1 | Demographics - All Included Population |
|---|---|
| Listing 16.2.4.2 | Magnetic Field in Tesla - All Included Population |
| Listing 16.2.4.3 | Current Renal Status - All Included Population |
| Listing 16.2.4.4 | Risk Factors and Medical History - All Included Population |
| Listing 16.2.4.5 | Previous Examinations with GBCA - All Included Population |

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

| Listing 16.2.4.6 | Recent Surgery - All Included Population |
|---|---|
| Listing 16.2.4.7 | Concomitant Medications - All Included Population |
| Listing 16.2.4.8 | Indication of Current MRI Examination - All Included Population |
| Listing 16.2.4.9 | Premedication - All Included Population |

# 6.3.5. Compliance and/or Drug Concentration Data

(Section 16.2.5 of ICH report)

Listing 16.2.5.1 DOTAREM® Administration - All Included Population

#### 6.3.6. Individual Efficacy Response Data

(Section 16.2.6 of ICH report)

Listing 16.2.6.1 Overall Quality of Images and Diagnostic Quality - All Included Population

#### 6.3.7. Adverse Event Listings

(Section 16.2.7 of ICH report)

Listing 16.2.7.1 Adverse Events - All Included Population

#### 6.3.8. Listing of Individual Laboratory Measurements

(Section 16.2.8 of ICH report)

Listing 16.2.8.1 Renal Status during Follow-up Period - All Included Population

#### 6.3.9. Vital signs, Physical Findings and Other Observations Related to Safety

(Section 16.2.9 of ICH report)

| Listing 16.2.9.1 | Nephrogenic Systemic Fibrosis Suspicion/Diagnosis - All Included Population |
|---|---|
| Listing 16.2.9.2 | Medical Events during Follow-up Period except MRI Examination - All Included Population |
| Listing 16.2.9.3 | MRI examination during Follow-up Period - All Included Population |

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

# 7. SHELLS FOR TABLES, FIGURES AND LISTINGS

All outputs will be produced using SAS® version 9.2.

The listings will include all patients and will be ordered by site and patient.

# 7.1. Clinical study report in-text tables, figures and listings

# 7.2. Contents of clinical study report section 14

Table 14.1.1.1 Patient Overall Disposition - All Included Population

| | | Total |
|---|---|---|
| | | (N=XXX) |
| Number of Patients not Prematurely | | xxx (xx.x%) |
| Withdrawn | | |
| Number of Patients Prematurely | | xxx (xx.x%) |
| Withdrawn | | ( ) |
| Reason of Withdrawal | Retraction of Patient Consent | xxx (xx.x%) |
| | Adverse Event | xxx (xx.x%) |
| | Patient Lost to Follow-up | xxx (xx.x%) |
| | Technical Incident | xxx (xx.x%) |
| | Death | xxx (xx.x%) |
| | Medical Decision | xxx (xx.x%) |
| | Other | xxx (xx.x%) |

%: (n row / N included) \* 100. Source: Listing 16.2.1.2.

Table 14.1.1.2 Disposition by Visit - All Included Population

| | General<br>Questionnaire | Follow-up 1<br>(N=XXX) | Follow-up 2<br>(N=XXX) | Follow-up 3<br>(N=XXX) | At Least<br>One Follow- |
|---|---|---|---|---|---|
| | (N=XXX) | | | | up Visit |
| Number of Patients | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

%: (n row / N included) \* 100. Source: Listing 16.2.1.1.

Table 14.1.1.3 Disposition by Site - All Included Population

| | | Total<br>(N=XXX) |
|-----------|---------|------------------|
| Argentina | Site 29 | xxx (xx.x%) |
| | Site 30 | xxx (xx.x%) |
| | Site 31 | xxx (xx.x%) |
| Belgium | Site 1 | xxx (xx.x%) |

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

| | | Total<br>(N=XXX) |
|--------------------------|---------|------------------|
| | Site 2 | xxx (xx.x%) |
| | Site 28 | xxx (xx.x%) |
| Brazil | Site 3 | xxx (xx.x%) |
| Columbia | Site 32 | xxx (xx.x%) |
| | Site 33 | xxx (xx.x%) |
| | Site 34 | xxx (xx.x%) |
| France | Site 6 | xxx (xx.x%) |
| | Site 26 | xxx (xx.x%) |
| Germany | Site 8 | xxx (xx.x%) |
| · | Site 27 | xxx (xx.x%) |
| India | Site 10 | xxx (xx.x%) |
| Italy | Site 12 | xxx (xx.x%) |
| | Site 13 | xxx (xx.x%) |
| | Site 14 | xxx (xx.x%) |
| Korea | Site 15 | xxx (xx.x%) |
| | Site 16 | xxx (xx.x%) |
| | Site 17 | xxx (xx.x%) |
| | Site 18 | xxx (xx.x%) |
| Spain | Site 19 | xxx (xx.x%) |
| | Site 20 | xxx (xx.x%) |
| | Site 35 | xxx (xx.x%) |
| Turkey | Site 23 | xxx (xx.x%) |
| | Site 37 | xxx (xx.x%) |
| United Kingdom | Site 24 | xxx (xx.x%) |
| | Site 25 | xxx (xx.x%) |
| Uruguay | Site 36 | xxx (xx.x%) |
| United States of America | Site 38 | xxx (xx.x%) |
| | Site 39 | xxx (xx.x%) |

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

| | Total<br>(N=XXX) |
|---------|------------------|
| Site 40 | xxx (xx.x%) |
| Site 41 | xxx (xx.x%) |

%: (n row / N included) \* 100. Source: Listing 16.2.1.1.

Table 14.1.1.4 Centre Characteristics and Radiological Activities - All Centres

| | Radiological Activities - All Centres | Total<br>(N=XX) |
|---|---|---|
| Type of Centre | n | XX |
| | Private | xx (xx.x%) |
| | Public | xx (xx.x%) |
| | Other | xx (xx.x%) |
| | Missing (if applicable) | XX |
| Radiological Fields or Specialities* | Neurology | xx (xx.x%) |
| | Cardiology | xx (xx.x%) |
| | Peripheral Vascular | xx (xx.x%) |
| | Musculoskeletal | xx (xx.x%) |
| | Oncology | xx (xx.x%) |
| | Other | xx (xx.x%) |
| Number of MR Equipment | n | XX |
| | 1 | xx (xx.x%) |
| | 2 | xx (xx.x%) |
| | 3 | xx (xx.x%) |
| | 4 | xx (xx.x%) |
| | 5 | xx (xx.x%) |
| | Missing (if applicable) | XX |
| Number of MR Examinations/Week | n | XXX |
| | Mean (SD) | xx.x(xx.x) |
| | Median | XX |
| | Min; Max | xx;xx |
| | Missing (if applicable) | XX |
| Usual Practice in MR Units | | |
| Allergic History Assessment | n | XX |
| | Yes | xx (xx.x%) |
| | No | xx (xx.x%) |
| | Missing (if applicable) | XX |

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

| | | Total<br>(N=XX) |
|---|---|---|
| Creatinine Level Assessment | n | XX |
| | Yes | xx (xx.x%) |
| | No | xx (xx.x%) |
| | Missing (if applicable) | XX |
| Other Assessment | n | XX |
| | Yes | xx (xx.x% |
| | No | xx (xx.x% |
| | Missing (if applicable) | XX |
| Patient Consent Form Signature | n | xx |
| | Yes | xx (xx.x% |
| | No | xx (xx.x% |
| | Missing (if applicable) | XX |
| Duration of Follow-up After MR<br>Examination | n | xx |
| | < 30 min | xx (xx.x% |
| | Between 30 min and 1 hour | xx (xx.x% |
| | > 1 hour | xx (xx.x% |
| | Missing (if applicable) | XX |

MR: Magnetic Resonance.

Table 14.1.1.5 Magnetic Fields of MR Equipments - All MR Equipments

| Table 14.1.1.5 Wagnetic | Wagnetie Fields of Wik Equipments - An Wik Equipments | |
|---|---|---|
| | | Total<br>(N=XX) |
| Magnetic Fields | 1.5 | xx (xx.x%) |
| | 3.0 | xx (xx.x%) |
| | Missing (if applicable) | xx |

MR: Magnetic Resonance.

%: (n row / N MR equipment) \* 100.

Source: Listing 16.2.1.3.

Table 14.1.2.1 Protocol Deviations - All Included Population

| Tuble 1 1.11.2.1 Trottocol Be viations | Till illeraded i opulation |
|----------------------------------------|----------------------------|
| | Total |
| | (N=XXX) |
| At Least One Protocol Deviation | xxx (xx.x%) |
| Protocol Deviation 1 | xxx(xx.x%) |
| Protocol Deviation n | xxx (xx.x%) |

<sup>%: (</sup>n row / n non missing) \* 100, except for multiple answers %: (n row / N centre) \* 100.

<sup>\*</sup>As multiple radiological fields or specialities are possible, the sum of percentage could be greater than 100. Source: Listing 16.2.1.3.

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

%: (n row / N included) \* 100. Source: Listing 16.2.2.1.

Table 14.1.3.1 Analysis Data Populations - All Included Population

| Total |
|-------------|
| (N=XXX) |
| xxx (xx.x%) |
| xxx (xx.x%) |

%: (n row / N included) \* 100. Source: Listing 16.2.3.1.

| | | Total |
|---|---|---|
| | | (N=XXX) |
| Sex | n | XXX |
| | Male | xxx (xx.x%) |
| | Female | xxx (xx.x%) |
| | Missing (if applicable) | XX |
| Age (years) for Patients Older than<br>Two Years Old | n | xxx |
| | Mean (SD) | xx.x(xx.x) |
| | Median | XX |
| | Min; Max | xx;xx |
| | Missing (if applicable) | XX |
| Age (month) for Patients Younger than Two Years Old | n | XXX |
| | Mean (SD) | xx.x (xx.x) |
| | Median | XX |
| | Min; Max | xx;xx |
| | Missing (if applicable) | XX |
| Weight (kg) | n | XXX |
| | Mean (SD) | xx.x(xx.x) |
| | Median | XX |
| | Min; Max | xx;xx |
| | Missing (if applicable) | XX |
| Height (cm) | n | XXX |
| | Mean (SD) | xx.x (xx.x) |
| | Median | XX |

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

| | | Total |
|---|---|---|
| | | (N=XXX) |
| | Min ; Max | xx;xx |
| | Missing (if applicable) | XX |
| Body Mass Index (kg/m²) | n | XXX |
| | Mean (SD) | xx.xx (xx.xx) |
| | Median | xx.x |
| | Min; Max | xx.x; xx.x |
| | Missing (if applicable) | XX |
| Body Mass Index by Class | n | xxx |
| | $< 18.5 \text{ kg/m}^2$ | xxx (xx.x%) |
| | $\geq$ 18.5 and $\leq$ 25 kg/m <sup>2</sup> | xxx (xx.x%) |
| | $\geq$ 25 and $\leq$ 30 kg/m <sup>2</sup> | xxx (xx.x%) |
| | $\geq 30 \text{ kg/m}^2$ | xxx (xx.x%) |
| | Missing (if applicable) | XX |

SD: Standard Deviation.

%: (n row / n non missing) \* 100.

Source: Listing 16.2.4.1.

Table 14.1.4.1.2 Demographic Characteristics – Safety Population

Same as table 14.1.4.1.2

Table 14.1.4.2 Magnetic Field - Safety Population

| - | - | Total |
|------------------------|-------------------------|-------------|
| | | (N=XXX) |
| Magnetic Field (Tesla) | n | XXX |
| | 1.5 | xxx (xx.x%) |
| | 3 | xxx (xx.x%) |
| | Missing (if applicable) | XX |

%: (n row / n non missing) \* 100. Source: Listing 16.2.4.2.

| Table 14.1.4.3 Current Renal Status - S | Safety Population | |
|---|---|---|
| | | Total |
| | | (N=XXX) |
| Intensity of Impaired Renal Function | n | XXX |
| | Moderate | xxx (xx.x%) |
| | Severe | xxx (xx.x%) |
| | End Stage Renal Insufficiency or Dialysis | xxx (xx.x%) |

CONFIDENTIAL

FORM

F015830-01

STATISTICAL ANALYSIS PLAN N° DGD-55-003

VERSION N° 2 DATED: 26 FEBRUARY 2018

(REF 1011622)

Page 30 / 49

| | | Total |
|---|---|---|
| | | (N=XXX) |
| | Kidney Transplantation | xxx (xx.x%) |
| | Missing (if applicable) | XX |
| If End Stage Renal Insufficiency or Dialysis, Specify | n | xxx |
| | Hemodialysis | xxx (xx.x%) |
| | Peritoneal Dialysis | xxx (xx.x%) |
| | Missing (if applicable) | XX |
| Most Recent Serum Creatinine (μmol/L) | n<br>No. (CD) | XXX |
| | Mean (SD) | xx.xx (xx.xx) |
| | Median | XX.X |
| | Min; Max | XX.X; XX.X |
| | Missing (if applicable) | XX |
| Estimated Creatinine Clearance (mL/min) for Patients Younger than 2 Years Old | | xxx (xx.x%) |
| If Yes, Estimated | n | xx |
| | Mean (SD) | xx.xx (xx.xx) |
| | Median | XX.X |
| | Min; Max | xx.x; xx.x |
| | Missing (if applicable) | xx |
| eGFR (mL/min/1.73 m²) for Patients<br>Older than 2 Years Old | | xxx (xx.x%) |
| If Yes, eGFR | n | xx |
| | Mean (SD) | xx.xx (xx.xx) |
| | Median | XX.X |
| | Min; Max | xx.x; xx.x |
| | Missing (if applicable) | XX |

eGFR: Estimated Glomerular Filtration Rate.

Source: Listing 16.2.4.3.

SD: Standard Deviation.

<sup>%: (</sup>n row / n non missing) \* 100, except for Estimated Creatinine Clearance and eGFR variables %: (n row / N safety population) \* 100.

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

Table 14.1.4.4 Pre-existing Risk Factor and Medical History - Safety Population

| | | Total |
|---|---|---|
| | | (N=XXX) |
| Liver Disorder | | xxx (xx.x%) |
| Allergies | | xxx (xx.x%) |
| Previous Reaction to Contrast Agents | | xxx (xx.x%) |
| | GBCA | xxx (xx.x%) |
| | Iodinated Contrast Agent | xxx (xx.x%) |
| Bronchial Asthma | | xxx (xx.x%) |
| Hypertension | | xxx (xx.x%) |
| Heart Insufficiency | | xxx (xx.x%) |
| | NYHA Class I | xxx (xx.x%) |
| | NYHA Class II | xxx (xx.x%) |
| | NYHA Class III | xxx (xx.x%) |
| | NYHA Class IV | xxx (xx.x%) |
| Other Cardiovascular Disease | | xxx (xx.x%) |
| Diabetes Mellitus | | xxx (xx.x%) |
| | Type I | xxx (xx.x%) |
| | Type II | xxx (xx.x%) |
| Proteinuria | | xxx (xx.x%) |
| Nervous System Disorders | | xxx (xx.x%) |
| At Risk Treatments | | xxx (xx.x%) |
| | Beta-Blockers | xxx (xx.x%) |
| | Interleukine2 | xxx (xx.x%) |
| | Other | xxx (xx.x%) |
| Hypothyroidism | | xxx (xx.x%) |
| History of Deep Venous Thrombosis | | xxx (xx.x%) |
| Erythropoietin | | xxx (xx.x%) |
| Acidosis | | xxx (xx.x%) |
| Hyperphosphatemia | | xxx (xx.x%) |
| Abnormal Ca <sup>++</sup> Level | | xxx (xx.x%) |
| High Serum Ferritin Level | | xxx (xx.x%) |

GBCA: Gadolinium based Contrast Agent; NYHA: New York Heart Classification.

Source: Listing 16.2.4.4.

Table 14.1.4.5 Previous Examinations with GBCA - Safety Population

| 1 4010 14.1.4.3 | Ticvious Ex | animations with ODCA | - Saicty I opulation |
|-----------------|-------------|----------------------|----------------------|
| | | | Total |
| | | | (N=XXX) |
| Previous Exami | nation | n | XXX |
| | | Yes | xxx (xx.x%) |
| | | No | xxx (xx.x%) |

<sup>%: (</sup>n row / N safety population) \* 100.

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

| | | Total |
|---------|-------------------------|-------------|
| | | (N=XXX) |
| | Missing (if applicable) | XX |
| If Yes* | Gadobutrol | xxx (xx.x%) |
| | Gadoterate Meglumine | xxx (xx.x%) |
| | ••• | |
| | Without Contrast | xxx (xx.x%) |
| | Missing | xxx (xx.x%) |

GBCA: Gadolinium based Contrast Agent.

Table 14.1.4.6 Recent Surgery - Safety Population

| | | Total |
|-----------------------------|-------------------------|-------------|
| | | (N=XXX) |
| At Least One Recent Surgery | n | XXX |
| | Yes | xxx (xx.x%) |
| | No | xxx (xx.x%) |
| | Missing (if applicable) | XX |

<sup>%: (</sup>n row / n non missing) \* 100.

Source: Listing 16.2.4.6.

Table 14.1.4.7 Concomitant Medications - Safety Population

| | | Total |
|-------------------------------------|-------------------------|-------------|
| | | (N=XXX) |
| At Least One Concomitant Medication | n | XXX |
| | Yes | xxx (xx.x%) |
| | No | xxx (xx.x%) |
| | Missing (if applicable) | XX |

<sup>%: (</sup>n row / n non missing) \* 100.

Source: Listing 16.2.4.7.

Table 14.1.4.8 Indication of MRI Examination - Safety Population

| | | Total |
|------------------------|-------------|-------------|
| | | (N=XXX) |
| Central Nervous System | | xxx (xx.x%) |
| | Head/Neck | xxx (xx.x%) |
| | Brain | xxx (xx.x%) |
| | Spinal Cord | xxx (xx.x%) |
| Whole Body | | xxx (xx.x%) |
| | Liver | xxx (xx.x%) |
| | Kidney | xxx (xx.x%) |

<sup>%: (</sup>n row / n with previous examination) \* 100, except for multiple answers %: (n row / n with previous examination) \* 100. \*As multiple examinations with various GBCA are possible, the sum of percentage could be greater than 100. Source: Listing 16.2.4.5.

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

| | | Total |
|------------------------------|--------------|-------------|
| | | (N=XXX) |
| | Pancreas | xxx (xx.x%) |
| | Pelvis | xxx (xx.x%) |
| Other Cardiovascular Disease | | xxx (xx.x%) |
| | Lung | xxx (xx.x%) |
| | Heart | xxx (xx.x%) |
| | Breast | xxx (xx.x%) |
| Musculoskeletal System | | xxx (xx.x%) |
| | Bones/Joints | xxx (xx.x%) |
| | Soft Tissue | xxx (xx.x%) |
| Angiography | | xxx (xx.x%) |
| | Carotids | xxx (xx.x%) |
| | Renal | xxx (xx.x%) |
| | Aorto Iliac | xxx (xx.x%) |
| | Calf | xxx (xx.x%) |
| | Other | xxx (xx.x%) |
| Other | | xxx (xx.x%) |

MRI: Magnetic Resonance Imaging. %: (n row / N safety population) \* 100. Source: Listing 16.2.4.8.

Table 14.1.4.9 Premedications - Safety Population

| | | Total |
|----------------------------|-------------------------|-------------|
| | | (N=XXX) |
| At Least One Premedication | n | XXX |
| | Yes | xxx (xx.x%) |
| | No | xxx (xx.x%) |
| | Missing (if applicable) | XX |

%: (n row / n non missing) \* 100. Source: Listing 16.2.4.9.

Table 14.2.2.1 Overall Quality of Images - Efficacy Population

| 1 4010 14.2.2.1 | Overall Quality of illiages | Differency i opulation | |
|---|---|---|---|
| | | | Total |
| | | | (N=XXX) |
| Image Quality | | n | XXX |
| | | Very Good | xxx (xx.x%) |
| | | Good | xxx (xx.x%) |
| | | Fair | xxx (xx.x%) |
| | | Poor | xxx (xx.x%) |
| | | Very Poor | xxx (xx.x%) |
| | | Missing (if applicable) | XX |

<sup>%: (</sup>n row / n non missing) \* 100.

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

Source: Listing 16.2.6.1.

Table 14.2.2.2 Diagnostic Quality - Efficacy Population

| | | Total<br>(N=XXX) |
|----------------|-------------------------|------------------|
| Diagnosis | n | xxx |
| | Yes | xxx (xx.x%) |
| | No | xxx (xx.x%) |
| | Missing (if applicable) | XX |
| If No, Reason* | Technical Problem | xxx (xx.x%) |
| | Anxious Patient | xxx (xx.x%) |
| | Other | xxx (xx.x%) |

<sup>%: (</sup>n row / n non missing) \* 100, except for multiple answers %: (n row / n with no diagnosis) \* 100. \*As multiple reasons are possible, the sum of percentage could be greater than 100.

Source: Listing 16.2.6.1.

Table 14.3.1.1 DOTAREM® Administration at Inclusion Visit - Safety Population

| | | Total |
|-----------------------------|-------------------------|---------------|
| | | (N=XXX) |
| Total Volume Injected (mL) | n | XXX |
| | Mean (SD) | xx.xx (xx.xx) |
| | Median | XX.X |
| | Min; Max | xx.x; xx.x |
| | Missing (if applicable) | XX |
| Total Dose Injected (mL/kg) | n | XXX |
| | Mean (SD) | xx.xx (xx.xx) |
| | Median | XX.X |
| | Min; Max | xx.x; xx.x |
| | Missing (if applicable) | XX |
| Type of Injection | n | XXX |
| | Manual | xxx (xx.x%) |
| | Automatic | xxx (xx.x%) |
| | Missing (if applicable) | XX |
| Number of Injections | n | XXX |
| | 1 | xxx (xx.x%) |
| | 2 | xxx (xx.x%) |
| | Missing (if applicable) | XX |
| Nature of Package | n | XXX |

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

| | | Total |
|-----------------------------------|----------------------------|-------------|
| | | (N=XXX) |
| | Vial | xxx (xx.x%) |
| | Pre-Filed Syringe | xxx (xx.x%) |
| | Vial and Pre-Filed Syringe | xxx (xx.x%) |
| | Missing (if applicable) | XX |
| Volume of Vial (mL) | n | XXX |
| | 5 mL | xxx (xx.x%) |
| | 10 mL | xxx (xx.x%) |
| | 15 mL | xxx (xx.x%) |
| | 20 mL | xxx (xx.x%) |
| | 60 mL | xxx (xx.x%) |
| | 100 mL | xxx (xx.x%) |
| | Missing (if applicable) | XX |
| Volume of Pre-filled Syringe (mL) | n | XXX |
| | 10 mL | xxx (xx.x%) |
| | 15 mL | xxx (xx.x%) |
| | 20 mL | xxx (xx.x%) |
| | Missing (if applicable) | XX |

SD: Standard Deviation. %: (n row / n non missing) \* 100.

Source: Listing 16.2.5.1.

Table 14.3.2.1 Suspected NSF - Safety Population

| | | Total |
|----------------------------|-------------------------|-------------|
| | | (N=XXX) |
| Suspicion of NSF | n | XXX |
| | Yes | xxx (xx.x%) |
| | No | xxx (xx.x%) |
| | Missing (if applicable) | xx |
| If Yes, | | |
| Skin* | Burning and Itching | xxx (xx.x%) |
| | Darkened Patches | xxx (xx.x%) |
| | Painful Skin Swelling | xxx (xx.x%) |
| Eyes* | Yellow Raised Spots | xxx (xx.x%) |
| Bones, Joints and Muscles* | Joint Stiffness | xxx (xx.x%) |
| | Limited Range of Motion | xxx (xx.x%) |

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

| | | Total |
|--------------------|----------------------------------|-------------|
| | | (N=XXX) |
| | Deep Pain | xxx (xx.x%) |
| | Muscle Weakness | xxx (xx.x%) |
| | Calcification of the Soft Tissue | xxx (xx.x%) |
| Systemic Fibrosis* | Fibrosis | xxx (xx.x%) |

NSF: Nephrogenic Systemic Fibrosis.

Table 14.3.2.2 Confirmatory Biopsy and Final Diagnosis - Safety Population - Patient with Suspicion of NSF

| | | Total |
|--------------------------------|-------------------------|-------------|
| | | (N=XXX) |
| Confirmatory Biopsy | n | XXX |
| | Yes | xxx (xx.x%) |
| | No | xxx (xx.x%) |
| | Missing (if applicable) | XX |
| If Yes, Final Diagnosis of NSF | n | XXX |
| | Yes | xxx (xx.x%) |
| | No | xxx (xx.x%) |
| | Missing (if applicable) | XX |

NSF: Nephrogenic Systemic Fibrosis.

Table 14.3.3.1 Overall Safety Summary - Safety Population

| | <b>Patients</b> | AEs |
|------------------------------------------------------|-----------------|-----|
| At Least One Adverse Event (AE) | xxx (xx.x%) | XXX |
| Distribution of AE | | |
| - 0 | xxx (xx.x%) | - |
| - 1 | xxx (xx.x%) | - |
| - 2 | xxx (xx.x%) | - |
| - 3 or more | xxx (xx.x%) | - |
| - Missing (if applicable) | XXX | - |
| At least one Treatment-Emergent Adverse Event (TEAE) | xxx (xx.x%) | XXX |
| At least one Serious Adverse Event (SAE) | xxx (xx.x%) | XXX |
| - Death | xxx (xx.x%) | xxx |
| - Life-threatening | xxx (xx.x%) | XXX |
| - Hospitalisation of Prolongation of Hospitalisation | xxx (xx.x%) | XXX |
| - Persistent or Significant Disability or Incapacity | xxx (xx.x%) | XXX |
| - Congenital Abnormality or Birth Defect | xxx (xx.x%) | XXX |
| - Medically Important | xxx (xx.x%) | XXX |

<sup>%: (</sup>n row / n non missing) \* 100, except for multiple answers %: (n row / n with suspicion of NSF) \* 100.

<sup>\*</sup>As the suspicion of NSF can be based on multiple topics, the sum of percentage could be greater than 100. Source: Listing 16.2.9.1.

<sup>%: (</sup>n row / n non missing) \* 100, except for Final Diagnosis of NSF %: (n row / n with confirmatory biopsy) \* 100. Source: Listing 16.2.9.1.
|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

| | <b>Patients</b> | AEs |
|---|---|---|
| - Missing (if applicable) | XXX | XXX |
| Intensity: At Least One AE: | | |
| - Mild | xxx (xx.x%) | XXX |
| - Moderate | xxx (xx.x%) | XXX |
| - Severe | xxx (xx.x%) | XXX |
| - Missing (if applicable) | XXX | XXX |
| Outcome: At Least One AE: | | |
| - Recovered | xxx (xx.x%) | XXX |
| - Not yet Recovered | xxx (xx.x%) | XXX |
| - Unknown | xxx (xx.x%) | XXX |
| - Missing (if applicable) | XXX | XXX |
| At Least One AE Requiring an Administration of Concomitant Drug | xxx (xx.x%) | XXX |

MedDRA dictionary version 16.0.

%: (n row / N safety population) \* 100.

Source: Listing 16.2.7.1.

Table 14.3.3.2 Treatment Emergent Adverse Events - Overall Summary - Safety Population

Same as table 14.3.3.1

Table 14.3.3.3 Pre-injection Adverse Events by Primary System Organ Class and Preferred Term - Safety Population

| | Total<br>(N=xxx) |
|-------------------|------------------|
| At Least One TEAE | xxx (xx.x%) |
| SOC 1 | xxx (xx.x%) |
| - PT 1 | xxx (xx.x%) |
| - PT 2 | xxx (xx.x%) |
| ••• | |
| SOC 1 | xxx (xx.x%) |
| - PT 1 | xxx (xx.x%) |
| - PT 2 | xxx (xx.x%) |

TEAE: Treatment Emergent Adverse Event.

MedDRA dictionary version 16.0.

%: (n row / N safety population) \* 100.

Source: Listing 16.2.7.1.

Table 14.3.3.4 Treatment Emergent Adverse Events by Primary System Organ Class and Preferred Term - Safety Population

Same as table 14.3.3.3

Table 14.3.3.5 Serious Treatment Emergent Adverse Events by Primary System Organ Class and Preferred Term - Safety Population

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

Same as table 14.3.3.3

Table 14.3.3.6 Treatment Emergent Adverse Events with Relationship to DOTAREM® by Primary System Organ Class and Preferred Term - Safety Population

Same as table 14.3.3.3

Table 14.3.3.7 Listing of Deaths - Safety Population

| | Primary System Organ<br>Class<br><sup>r</sup> Preferred Term<br>Description | Start Date & Time/ | Seriousness/<br>Outcome | Intensity / Relationship to DOTAREM® | Administration<br>of Concomitant<br>Drug | |
|---|---|---|---|---|---|---|
| xxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xmm/dd/yyyy<br>hh:mm/ | Death/ | xxxxxxxxxxxx/ | xxxxxxxxxxxx/ | mm/dd/yyyy<br>hh:mm |
| | xxxxxxxxxxxxxxxxxx | mm/dd/yyyy<br>hh:mm | Life-<br>threatening | xxxxxxxxxxxx | xYes/No/ | |
| | xxxxxxxxxxxxxxxxxx | XXXX | | | Yes/No | |

Etc.

MRI: Magnetic Resonance Imaging. MedDRA dictionary version 16.0. Source: Listing 16.2.7.1.

Listing of Serious Adverse Events - Safety Population Table 14.3.3.8

Same as table 14.3.3.7

Table 14.3.4.1 Renal Status during Follow-up Period - Safety Population

| | | Follow-up 1 | Follow-up 2 | Follow-up 3 |
|---|---|---|---|---|
| | | (N=XXX) | (N=XXX) | (N=XXX) |
| Serum Creatinine (Raw<br>Data) | n | xxx | xxx | xxx |
| | Mean (SD) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| | Median | xx.x | XX.X | xx.x |
| | Min; Max | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x |
| | Missing (if applicable) | XX | XX | XX |
| Serum Creatinine (Change from Baseline) | n | xxx | XXX | XXX |
| | Mean (SD) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min; Max | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x |
| | Missing (if applicable) | XX | XX | XX |

SD: Standard Deviation. Source: Listing 16.2.8.1.

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

Table 14.3.5.1 Medical Events except MRI Examination during Follow-up Period - Safety Population

| | | Follow-up 1 Follow-up 2 Follo | | |
|---|---|---|---|---|
| | | (N=XXX) | (N=XXX) | (N=XXX) |
| Surgery | n | xxx | XXX | xxx |
| | Yes | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | No | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Missing (if applicable) | XX | XX | XX |
| Pro-Inflammatory<br>Syndrom | n | xxx | XXX | xxx |
| | Yes | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | No | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Missing (if applicable) | XX | XX | XX |
| Hepato-Renal Syndrom | n | XXX | XXX | xxx |
| | Yes | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | No | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Missing (if applicable) | XX | XX | XX |
| Liver Transplant | n | XXX | XXX | XXX |
| | Yes | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | No | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Missing (if applicable) | XX | XX | xx |
| Other | n | xxx | xxx | xxx |
| | Yes | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | No | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Missing (if applicable) | XX | XX | XX |

MRI: Magnetic Resonance Imaging.

%: (n row / n non missing) \* 100.

Source: Listing 16.2.9.2.

Table 14.3.5.2 Contrast Media for MRI Examination during Follow-up Period - Safety Population

| | | Follow-up 1 | Follow-up 2 | Follow-up 3 |
|---|---|---|---|---|
| | | (N=XXX) | (N=XXX) | (N=XXX) |
| MRI Examination | n | XXX | xxx | xxx |
| | Yes | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | No | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Missing (if applicable) | XX | XX | XX |
| If Yes* | Gadobutrol | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

| | Follow-up 1 | Follow-up 2 | Follow-up 3 |
|----------------------|-------------|-------------|-------------|
| | (N=XXX) | (N=XXX) | (N=XXX) |
| Meglumine Gadoterate | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Without Contrast | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Missing | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

MRI: Magnetic Resonance Imaging.

Table 14.3.5.3 Medical Events except MRI Examination during Follow-up Period by Primary System Organ Class and Preferred Term - Safety Population

| | | Follow-up 1 | Follow-up 2 | Follow-up 3 |
|---------|----------------------|-------------|-------------|-------------|
| | | (N=XXX) | (N=XXX) | (N=XXX) |
| Surgery | At Least One Surgery | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | SOC 1 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | - PT 1 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | - PT 2 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

**Pro-Inflammatory Process** 

Etc...

MedDRA dictionary version 16.0. %: (n row / N column) \* 100. Source: Listing 16.2.9.2.

<sup>%: (</sup>n row / n non missing) \* 100, except for multiple answers %: (n row / n with MRI examination) \* 100.

<sup>\*</sup>As multiple examinations with various GBCA are possible for each visit, the sum of percentage could be greater than 100. Source: Listing 16.2.9.3.

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

## 7.3. Contents of clinical study report section 16.2

Listing 16.2.1.1 Visit Dates - All Included Population

| Patient # | Country | Centre # | Date of MRI | Date of | Date of | Date of |
|---|---|---|---|---|---|---|
| | | | Examination | Follow-up 1 | Follow-up 2 | Follow-up 3 |

MRI: Magnetic Resonance Imaging.

Listing 16.2.1.2 Premature Withdrawal - All Included Population

| Patient # | Date of Withdrawal | Premature Withdrawal | Who Decided the Withdrawal | Reason of Withdrawal |
|---|---|---|---|---|
|---|---|---|---|---|

Listing 16.2.1.3 Centre Characteristics and Radiological Activities

| Centre # | Type | Radiological Fields or Specialities | Number of MR<br>Equipments | Magnetic<br>Field | Number of MR<br>Examinations/Week | <b>Usual Practices in MR Units</b> | Duration of FU After MR<br>Examination |
|---|---|---|---|---|---|---|---|
| 01 | Public | Neurology/Cardiology | 2 | 1.5/1.5 | 156 | Allergic History assessment/ Other<br>Assessment: RAUPSE | < 30 min |

MR: Magnetic Resonance; FU: Follow-Up.

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

Listing 16.2.2.1 Protocol Deviations - All Included Population

Patient # Deviation Term Deviation Code

Listing 16.2.3.1 Analysis Data Populations - All Included Population

Patient # Efficacy Population Safety Population

Listing 16.2.4.1 Demographics - All Included Population

| Patient # | Population | Age | Age | Height (cm) | Weight (kg) | BMI | Sex |
|---|---|---|---|---|---|---|---|
| | Flag | (years) | (months) | | | $(kg/m^2)$ | |

AIP: All Included Population; EP: Efficacy Population; SP: Safety Population; BMI: Body Mass Index.

Listing 16.2.4.2 Magnetic Field in Tesla - All Included Population

Patient # Population Magnetic Field Flag (Tesla)

AIP: All Included Population ; EP: Efficacy Population ; SP: Safety Population.

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

Listing 16.2.4.3 Current Renal Status - All Included Population

| Patient # | Population | Renal | Most recent Serum | Most recent | Unit | Date | <b>Estimated Creatinine</b> | eGFR |
|---|---|---|---|---|---|---|---|---|
| | Flag | Function | Creatinine | Serum Creatinine | | | Clearance (mL/min) | (mL/min/1.73m2) |
| | | | (umol/L) | (entered) | | | | |

AIP: All Included Population; EP: Efficacy Population; SP: Safety Population; eGFR: estimated Glomerular Filtration Rate.

Listing 16.2.4.4 Risk Factors and Patient History - All Included Population

| Patient # | Population | Risk | Result | Specify |
|-----------|------------|--------|--------|---------|
| | Flag | Factor | | |

AIP: All Included Population ; EP: Efficacy Population ; SP: Safety Population.

Listing 16.2.4.5 Previous Examinations with GBCA - All Included Population

| Patient<br># | Population<br>Flag | Previous<br>Examination | Number of Examination | Examination<br>Date | <b>Product Class</b> | Product Name | Volume<br>Administered<br>(mL) |
|---|---|---|---|---|---|---|---|
| 001 | AIP/EP/SP | No | | | | | |
| 002 | | Yes | 3 | 13MAR2002 | Gadobutrol | GADOVIST® | 10 |
| 002 | | Yes | 3 | 15APR2003 | Gadoterate Meglumine | <b>DOTAREM®</b> | 20 |

AIP: All Included Population; EP: Efficacy Population; SP: Safety Population.

# CONFIDENTIAL STATISTICAL ANALYSIS PLAN N° DGD-55-003 VERSION N° 2 DATED: 26 FEBRUARY 2018 (REF 1011622) F015830-01 F015830-01

Listing 16.2.4.6 Recent Surgery - All Included Population

| Patient # | Population<br>Flag | Surgery | Description |
|-----------|--------------------|---------|-------------|
| 001 | AIP/EP/SP | Yes | |

AIP: All Included Population; EP: Efficacy Population; SP: Safety Population.

Listing 16.2.4.7 Concomitant Medications - All Included Population

| Patient # | Population<br>Flag | Concomitant Treatment |
|-----------|--------------------|-----------------------|
| 001 | AIP/EP/SP | XXXX |

AIP: All Included Population; EP: Efficacy Population; SP: Safety Population.

Listing 16.2.4.8 Indication of Current MRI Examination - All Included Population

| Patient # | Population<br>Flag | Classification | Sub Classification | Specify |
|---|---|---|---|---|
| 001 | AIP/EP/SP | | | |

AIP: All Included Population; EP: Efficacy Population; SP: Safety Population.

# CONFIDENTIAL STATISTICAL ANALYSIS PLAN N° DGD-55-003 VERSION N° 2 DATED: 26 FEBRUARY 2018 (REF 1011622) F015830-01 F015830-01

Listing 16.2.4.9 Premedication - All Included Population

| Patient # | Population<br>Flag | Premedication | Specify |
|-----------|--------------------|---------------|---------|
| 001 | AIP/EP/SP | Yes | XXXXX |

AIP: All Included Population; EP: Efficacy Population; SP: Safety Population.

Listing 16.2.5.1 DOTAREM® Administration – All Included Population

| Patient<br># | Population<br>Flag | Total Volume (mL) | Total Dose (mL/kg) | Type of Injection | Number of<br>Injection | Nature of<br>Package | Volume<br>of Vial | Volume of Pre-<br>filled Syringe |
|---|---|---|---|---|---|---|---|---|
| 001 | AIP/EP/SP | | | | | | | |

AIP: All Included Population; EP: Efficacy Population; SP: Safety Population.

Listing 16.2.6.1 Overall Quality of Images and Diagnostic Quality- All Included Population

| Patient # | Population Flag | Image Quality | Comment | Diagnosis | Specify | Reason |
|---|---|---|---|---|---|---|
| 001 | AIP/EP/SP | Fair | XXXXX | Yes | XXX | |
| 001 | AIP/EP/SP | | | No | | XXXX |

AIP: All Included Population; EP: Efficacy Population; SP: Safety Population.

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

Listing 16.2.7.1 Adverse Events - All Included Population

| Patient<br># | Population<br>Flag | Primary System Organ Class<br>Preferred Term<br>Nature of the Event | Start Date | Seriousness/<br>Outcome | Intensity / Relationship to DOTAREM® | Administration of Concomitant Drug | Date of MRI<br>Examination with<br>DOTAREM® |
|---|---|---|---|---|---|---|---|
| XXXX | | xxxxxxxxxxxxxxxxx | mm/dd/yyyy | Yes:Death/ not y recovered | vet Moderate/Not related | Yes :xxxxxxx | mm/dd/yyyy |
| | | xxxxxxxxxxxxxxxx | mm/dd/yyyy | No/recovered | Mild/unknown | No | |

### Etc.

AIP: All Included Population ; EP: Efficacy Population ; SP: Safety Population ; MRI: Magnetic Resonance Imaging. MedDRA dictionary version 16.0.

Listing 16.2.8.1 Renal Status during Follow-up Period - All Included Population

| Patient # | Population<br>Flag | Date of MRI<br>Examination | Follow-up<br>Visit | Date of Last<br>Renal Function | Serum<br>Creatinine | Serum<br>Creatinine | Unit |
|---|---|---|---|---|---|---|---|
| | | with<br>DOTAREM® | | Assessment | (umol/L) | (Entered) | |

AIP: All Included Population; EP: Efficacy Population; SP: Safety Population; MRI: Magnetic Resonance Imaging.

Listing 16.2.9.1 Nephrogenic Systemic Fibrosis Suspicion/Diagnosis - All Included Population

| Patient # Po | opulation<br>Flag | Date of MRI<br>Examination with<br>DOTAREM® | NSF<br>Suspicion | Source of Suspicion | Confirmatory<br>Biopsy | Specify if No | Date of the<br>Biopsy | Final Diagnosis<br>of NSF | Specify if No |
|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

AIP: All Included Population; EP: Efficacy Population; SP: Safety Population; MRI: Magnetic Resonance Imaging; NSF: Nephrogenic Systemic Fibrosis.

Listing 16.2.9.2 Medical Events during Follow-up Period except MRI examination - All Included Population

| Patient # | Population<br>Flag | Date of MRI<br>Examination with<br>DOTAREM® | Follow-up<br>Visit | Date of FU<br>Visit | Medical<br>Event<br>Category | Medical<br>Event Date | Primary System Organ Class<br>(Preferred Term)<br>[Description] | Medical Event<br>Specify |
|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|

AIP: All Included Population; EP: Efficacy Population; SP: Safety Population; MRI: Magnetic Resonance Imaging; FU: Follow-Up. MedDRA dictionary version 16.0.

Listing 16.2.9.3 MRI examination during Follow-up Period - All Included Population

| Patient # | Population | Follow-up | Date of FU | Product | Product | Product | Volume | Date |
|---|---|---|---|---|---|---|---|---|
| | Flag | Visit | Visit | ATC Name | Class | Name | Administered (mL) | |

AIP: All Included Population; EP: Efficacy Population; SP: Safety Population; ATC: Anatomical Therapeutic Chemical; FU: Follow-Up. WHO DD dictionary version 2015.

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

## 8. REFERENCES

[1] Iverson C, Flanagan A, Fontanarosa PB, et al American Medical Association Manual of Style: A Guide for authors and Editors.  $9^{th}$  ed

ICH-E3 Note for Guidance on Structure and Content of Clinical Study Reports

|-----------------------------------------|
| STATISTICAL ANALYSIS PLAN N° DGD-55-003 |
| (REF 1011622) |

## 9. APPENDICES